CLINICAL TRIAL: NCT04569227
Title: Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of EC-18 in Preventing the Progression of COVID-19 Infection to Severe Pneumonia or ARDS
Brief Title: Prevention of COVID-19 Infection to Severe Pneumonia or ARDS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Enzychem Lifesciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC-18-204
Record Dates: First submitted 2020-09-28; First posted 2020-09-29 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-04

CONDITIONS: Covid19 Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active EC-18 (Experimental)
  Interventions: Drug: EC-18
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EC-18 — 2000 mg PO daily
  Arms: Active EC-18
Drug: Placebo — PO daily
  Arms: Placebo

SUMMARY:
A trial of EC-18 in patients with mild/moderate pneumonia due to COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria:

  1. Male or female ≥18 years old
  2. Subjects with confirmed diagnoses of pneumonia caused by COVID-19 from:

     * RT-PCR or Abbott ID Now COVID-19 test
     * Chest X-ray or computed tomography (CT) scan (findings of the increased opacity on a chest X-ray, ground-glass opacity indicative of pneumonia on CT, opinion on consolidation, etc.)
  3. Those who can tolerate oral administration
  4. Those who do not need oxygen therapy or only need low-flow oxygen (at least 4L/min) but not requiring high-flow oxygen (higher than 4-6L/min) or non-invasive/invasive ventilation primarily according to the WHO guidance
  5. Those who are planned to be hospitalized or who are just hospitalized
  6. Those who have been fully explained about this clinical study and have voluntarily agreed to participate in this clinical study by signing the informed consent form (ICF)

Exclusion Criteria:

* Subjects cannot participate in this clinical study if they satisfy any of the following criteria:

  1. Those who are diagnosed with viral pneumonia caused by other than COVID-19 or bacterial pneumonia during the screening
  2. Patients with severe pneumonia according to the WHO guidance

     * Have fever or signs of respiratory infections and
     * Satisfy any one of the following conditions: Respiratory rate > 30 breaths/min, severe respiratory distress, or room air oxygen saturation (SpO2) ≤ 93%
  3. Patients with ARDS according to the WHO guidance
  4. Those who have past medical histories described below:

     * Those who have medical histories of human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS), or hepatitis B or C viral infection
     * Those who cannot have a CT test done due to allergy to contrast agents, etc.
  5. Those who have comorbidities/symptoms described below:

     * Those who have a history or evidence of another clinically significant condition that may pose risks to patient safety or interfere with the study procedures, assessments or completion as determined by the investigator
     * Those who have moderate or severe renal impairment (eGFR < 60 mL/min/1.73 m2)
     * Those who have moderate or severe hepatic impairment (Child-Pugh B or C, respectively)
  6. Patients who are being treated with corticosteroids or other immunosuppressants for asthma or autoimmune diseases at the entry of study are excluded, because these drugs counteract the action mechanism of EC-18 (PLAG).
  7. Those who have any abnormalities in laboratory tests described below:

     * Clinically significant liver function abnormality (Satisfy any one or more of the following):
     * Serum alanine aminotransferase (ALT) ≥ upper limit of normal (ULN) × 2.5
     * Serum aspartate aminotransferase (AST) ≥ ULN × 2.5
     * Serum total bilirubin ≥ ULN × 2.5
  8. Patients with uncontrolled diabetes (HbA1c > 7.0%)
  9. Those who have hypersensitivity reactions to the IP and its components
  10. Those who satisfy any of the descriptions below:

      * Pregnant or breastfeeding female subjects
      * Those who are planning on pregnancy or not using accepted contraception measures during the clinical study
  11. Those who have participated in other clinical studies to receive IPs or apply investigational medical devices within 1 month from the time of obtaining the informed consent
  12. Those who are considered to be ineligible to participate in the clinical study or have difficulty conducting this clinical study by the investigator
  13. Those subjects with Hb < lower limit of normal (LLN) for males and females
  14. Those subjects with a platelet count < LLN
  15. Those subjects with a WBC < LLN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients alive and free of respiratory failure through at Day 28 | 28 days

SECONDARY OUTCOMES:
Probability of progression of mild pneumonia patients to severe pneumonia or ARDS within 28 days | 28 days
Assessment of all-cause mortality | 28 days
Respiratory failure defined based on resource utilization requiring at least 1 of the following: | 28 days
  * Endotracheal intubation and mechanical ventilation
  * Oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates > 20L/min with a fraction of delivered oxygen ≥ 0.5)
  * Non-invasive positive pressure ventilation
  * Extracorporeal membrane oxygenation
Proportion of patients alive and free of invasive mechanical ventilation at a pre-specified timepoint | 28 days
Proportion of patients alive and discharged from the hospital at a pre-specified timepoint | 28 days
Lengths of ICU stay | 28 days
Lengths of alive and respiratory failure-free days | 28 days
Proportion of patients with objective measures of improvement (returning to room air) at time points (days 7, 14, and 28) | 7, 14, and 28 days
Confirmation of changes in subject's subjective clinical symptoms (e.g., patient questionnaire) | 28 days
  o Check for changes in symptoms on a daily basis for 28 days compared to the baseline at day 1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lincoln Medical Center, The Bronx, New York
  - Kent County Memorial Hospital, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: No